CLINICAL TRIAL: NCT07165704
Title: Community Galleries - Art and Children in Action: Protocol for a Cluster Non-Randomized Controlled Trial of an Art-Based Intervention to Promote Child Psychological Adjustment, Self-Concept and Quality of Life
Brief Title: Community Galleries - Art and Children in Action: Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associação para o Apoio à Integração Social e Comunitária (Other)
Collaborators: Fundação Caloust Gulbenkian (Unknown); Uppsala University (Other); Lusofona University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ESPACOT1220425
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Self-concept; Psychological Adjustment; Health Related Quality of Life
Keywords: Self-concept; Health-related quality of life; Quality-adjusted life years; Psychological adjustment; Arts-based intervention; Visual arts; Cost-utility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual Art Intervention (Experimental): The arts intervention will consist of two parts: (a) implementation of one-hour session of Visual Arts (e.g., painting, drawing, printing techniques exercises). (b) Children's final artistic products will be displayed in Community Galleries in their neighbourhood in an opening ceremony.
  Interventions: Other: Visual arts
- Waitlist Control (No Intervention)

INTERVENTIONS:
Other: Visual arts — The arts intervention will consist of two parts: (a) implementation of one-hour session of Visual Arts (e.g., painting, drawing, printing techniques exercises). The activities will be guided through a theme (Emotions), by a professional artist, to obtain a final individual artistic product. Peer contact, shared learning, and a feeling of community are all made possible by the group-based approach. This facilitator will offer assistance, motivation, and technical training as they lead participants through the creative process. Using narrative-building and dialogue-based methods, the artist will encourage children to share their stories, experiences, and perspectives, through art. (b) Children's final artistic products will be displayed in Community Galleries in their neighbourhood in an opening ceremony.
  Other Names: Community Galleries
  Arms: Visual Art Intervention

SUMMARY:
The goal of this trial is to evaluate whether a community-based visual arts intervention can improve self-concept, psychological adjustment, and health-related quality of life (HRQoL) in children aged between 6 and 12, from socioeconomically disadvantaged neighborhoods.

The main questions it aims to answer are:

* Does the intervention improve children's psychological adjustment, as the primary outcome?
* Does the intervention improve self-concept and health-related quality of life (HRQoL) as the secondary outcomes?
* Is the intervention cost-effective compared to the waitlist control?

Researchers will compare children receiving the visual arts intervention (intervention group) with children not receiving the intervention (waiting list control group) to see if the program leads to measurable improvements in psychological adjustment, self-concept, and health-related quality of life.

Participants will:

* Take part in one-hour weekly visual arts sessions for nine months, led by professional artists;
* Participate in community art exhibitions at the end of the program;
* Complete questionnaires on psychological adjustment, self-concept, HRQoL, and societal resource use at baseline and post-intervention;
* Teachers/technicians will complete questionnaires on children's psychological adjustment.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in elementary school and registered as a participant or student in one of the 10 schools or institutions, partners of the Community Galleries project.

Exclusion Criteria:

* Cognitive deficit, neurological disease or global developmental disorder

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total difficulties as assessed by The Strengths and Difficulties Questionnaire. | Baseline and 9 months
  The Strengths and Difficulties Questionnaire (SDQ) produces a total difficulties score ranging from 0 to 40, with higher scores indicating greater difficulties. It also comprises five subscales, each scored from 0 to 10: Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, Peer Relationship Problems, and Prosocial Behaviour (for which higher scores indicate more prosocial behaviours).

SECONDARY OUTCOMES:
Change from baseline of Self-concept as assed by The Self-Perception Profile for Children and the The Pictorial Scale of Perceived Competence and Social Acceptance for Young Children. | Baseline and 9 months
  This outcome is mesured with a) The Self-Perception Profile for Children (SPPC) produces domain-specific scores and a global self-worth score, each ranging from 1 (lowest perceived self-concept) to 4 (highest perceived self-concept). The scale includes six domains: Scholastic Competence, Social Acceptance, Athletic Competence, Physical Appearance, Behavioural Conduct, and Global Self-Worth. For children 7 years old and over; and b) The Pictorial Scale of Perceived Competence and Social Acceptance for Young Children produces scores for four domains: Cognitive Competence, Physical Competence, Peer Acceptance, and Maternal Acceptance, each ranging from 1 (lowest perceived competence or acceptance) to 4 (highest perceived competence or acceptance), for chindren under 7 years.
Quality-adjusted life years (QALY) gains from baseline as assed by the Child Health Utility 9 Dimensions. | Baseline and 9 months.
  To assess this outcome, the Child Health Utility 9 Dimensions is a health-related quality of life (HRQoL) measure designed for use in children. The CHU9D captures nine dimensions: worry, sadness, pain, tiredness, annoyance, schoolwork, sleep, routine, and activities. For each dimension, a five-level ordinal scale is used from 1 (no problems) to 5 (severe problems). Intended for use in cost-effectiveness evaluations of youth-focused treatment and assistance initiatives the instrument derives a single utility score of the health state experienced by the child from preference weights. CHU9D utility scores will be used to estimate QALYs (Quality Of Life in Years) for children over the study period using the area under the curve method. The range of utility scores is from 0 (where it will be equal to dead state) to 1 (where it will be in perfect health state), which is a part of cost-utility analysis, especially in economic evaluation.

OTHER OUTCOMES:
Change from baseline on children´s use of societal resources | Baseline and 9 Months
  A parent-reported resource use questionnaire will also be administered to collect information on children´s use of societal resources

CONTACTS AND LOCATIONS:
Overall Officials: Sandra P Henriques, Mastre, Principal Investigator — Associação Para o Apoio e Integração Social e Comunitária
Locations (10):
- Portugal (10):
  - Associação de Solidariedade da Zona das Fontainhas, Porto
  - Espaço Raíz, Porto
  - Escola do Parque Centro de Bem-estar Social Nossa Senhora do Socorro, Porto
  - A Associação de Promoção Social da População do Bairro do Aleixo, Porto
  - ASAS (Associação de Solidariedade e Ação Social de Ramalde), Porto
  - Paróquia de Nossa Senhora da Ajuda - Pasteleira, Porto
  - Escola Básica do Falcão, Porto
  - Centro Social do Lagarteiro, Porto
  - Escola Básica de Montebello, Porto
  - Escola Básica de São Roque da Lameira, Porto

IPD SHARING:
Plan to Share IPD: Undecided